CLINICAL TRIAL: NCT06907875
Title: A Phase 1/2 Open-label Dose-escalation Study to Evaluate the Safety, Tolerability, and Biological Activity of EPI-321, an AAVrh74-delivered Epigenetic Editing Therapy in Adult FSHD Patients
Brief Title: A First-in-human Study of EPI-321 in Facioscapulohumeral Muscular Dystrophy
Acronym: FSHD
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Epicrispr Biotechnologies, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: EPI-321-02
Record Dates: First submitted 2025-03-26; First posted 2025-04-02 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-05

CONDITIONS: Facioscapulohumeral Muscular Dystrophy
Keywords: Facioscapulohumeral Muscular Dystrophy; EPI-321; Muscular Dystrophy
MeSH Terms: conditions — Muscular Dystrophy, Facioscapulohumeral; Muscular Dystrophies

STUDY DESIGN:
Intervention Model Description: Dose escalation with two dose levels
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- EPI-321 Cohort 1 Single IV Dose (Experimental): Single IV infusion of a target dose of 2x10^13 vg/kg
  Interventions: Biological: EPI-321
- EPI-321 Cohort 2 Single IV Dose (Experimental): Single IV infusion of a target dose of 4x10^13 vg/kg
  Interventions: Biological: EPI-321

INTERVENTIONS:
Biological: EPI-321 — EPI-321 IV Infusion

SUMMARY:
The goal of this clinical trial is to learn how safe and tolerable EPI-321 is and whether there may be early signs it is working in male or female adult (18 to 75 years) participants with facioscapulohumeral muscular dystrophy (FSHD) Type 1 condition. The main questions it aims to answer are:

How safe is EPI-321 and how well can people handle it over time? How does EPI-321 interact with its target and does it show early signs of working?

Participants will receive a single dose of EPI-321 through a vein while being closely watched in a hospital and visit the clinic regularly for tests and checkups for about 5 years after getting EPI-321.

DETAILED DESCRIPTION:
EPI-321 is an investigational drug product comprising a recombinant adeno-associated viral vector, serotype rh74 (AAVrh74), for the delivery of genetic material encoding an epigenetic editor designed to address the root case of FSHD. AAVrh74 has been shown to transduce human skeletal muscle efficiently in the clinical experience. EPI-321's transgene product, a non-cutting, nuclease-dead mini, clustered regularly interspaced short palindromic repeat (CRISPR)-associated protein (dCasONYX) with fuse epigenetic modulators, is designed to selectively bind the D4Z4 repeat region via the accompanying guide RNA, methylate CpG groups within the region near the DUX4 gene on chromosome 4q35, and thus repress the expression of toxic DUX4 protein, ameliorating the downstream pathology that drives FSHD. As it is under a muscle-specific promoter, the dCasONYX-fused protein is expected to be preferentially and actively expressed in muscle tissue following a single intravenous (IV) dose.

EPI-321-02 clinical trial is an open label dose ascending study of EPI-321 for safety and tolerability to determine the best dose for a future trial of drug activity. Two dose levels will be evaluated. In addition, this study will collect secondary outcome data on muscle function, imaging characteristics, and other markers of disease activity at the baseline and throughout the study to assess their utility as measures of drug activity in a future clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Able and willing to provide informed consent
* Male or female 18 to 75 years of age
* Clinical diagnosis of FSHD with genetic Type 1
* FSHD Ricci clinical severity score 2 to 4 (on 5-point scale)
* Has adequate liver function
* Has adequate kidney function

Exclusion Criteria:

* Has an anti-AAVrh74 total binding antibody titer > 1:400
* Requires a walker or wheelchair for ambulation
* Pregnant and/or breastfeeding at baseline or is planning to become pregnant during the first 12 months following EPI-321 administration
* Has FSHD Type 2
* Has a concurrent or past medical conditions could jeopardize the safety of the participant

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-05-08 (Actual); Primary Completion 2031-03-31 (Estimated); Study Completion 2032-04-30 (Estimated)

PRIMARY OUTCOMES:
Frequency of AEs and EPI-321 Related Adverse Reactions and Serious Adverse Reactions | Baseline to up to 5 years.
  All AEs, regardless of assessed relatedness to EPI-321, will be collected from the time of informed consent signature until the end of study participation. The Investigator is responsible for assessing the severity of an AE according to the NCI-CTCAE version 5.0.

SECONDARY OUTCOMES:
Vector Copy Number | Baseline, 3 and 12 months
  Change in vector copy number (as measured by vg/dg) within skeletal muscle biopsies.
EPI-321 Cargo Transcriptional Activity | Baseline, 3 and 12 months
  Change in EPI-321 cargo transcriptional activity within skeletal muscle biopsies.
DUX4 Expression | Baseline, 3 and 12 months
  Change in the expression of DUX4 and downstream markers (DUX4 Composite Score) within skeletal muscle biopsies.
Methylation Status | Baseline, 3 and 12 months
  Change from baseline in the methylation status of the 4q35 D4Z4 region within skeletal muscle biopsies at 3 and 12 months.

CONTACTS AND LOCATIONS:
Locations (6):
- United States (4):
  - David Geffen School of Medicine at University of California, Los Angeles, Los Angeles, California
  - Rare Disease Research, Atlanta, Georgia
  - University of Massachusetts Chan Medical School, Worcester, Massachusetts
  - Utah Program for Inherited Neuromuscular Disorders - University of Utah, Salt Lake City, Utah
- Royal Alfred Hospital, Sydney, New South Wales, Australia
- Pacific Clinical Research Network, Auckland, New Zealand

IPD SHARING:
Plan to Share IPD: No